CLINICAL TRIAL: NCT00239226
Title: Investigational New Drug Application/ Investigational Device Exemption Information
Brief Title: Electrophysiologically Guided PAcing Site Selection Study
Acronym: EPASS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic BRC (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EPASS
Record Dates: First submitted 2005-10-13; First posted 2005-10-14 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2012-04

CONDITIONS: Sinus Arrhythmia; Atrial Fibrillation
Keywords: atrial fibrillation; interatrial septum; atrial pacing; symptomatic sinus node dysfunction,; pacemaker indication class I
MeSH Terms: conditions — Arrhythmia, Sinus; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1. IAS pacing - study group (Experimental): Patients were first submitted to electrophysiological study to assess Delta CTos > or < 50 ms. Then they were randomized to interatrial septum pacing od right atrial appendage. This arm (1) includes patients with Delta CTos >50 ms and randomized IAS pacing.
  IAS Pacing -Study Group: Patients with Delta CTos >50 ms (study group) at the electrophysiologic study and randomized Interatrial Septum Pacing
  Interventions: Procedure: IAS pacing - study group
- 2. IAS pacing-control group (Experimental): (Delta CTos<50ms)
  Patients were first submitted to electrophysiological study to assess Delta CTos > or < 50 ms. Then they were randomized to interatrial septum pacing od right atrial appendage. This arm (2) includes patients with Delta CTos <50 ms and randomized IAS pacing.
  IAS Pacing -Control Group: Patients with Delta CTos <50 ms (control group) at the electrophysiologic study and randomized Interatrial Septum Pacing
  Interventions: Procedure: IAS pacing control group
- 3. RAA Pacing - study group (Active Comparator): Patients were first submitted to electrophysiological study to assess Delta CTos > or < 50 ms. Then they were randomized to interatrial septum pacing od right atrial appendage. This arm (3) includes patients with Delta CTos >50 ms and randomized Right Atrial Appendage pacing.
  RAA Pacing -Study Group: Patients with Delta CTos >50 ms (study group) at the electrophysiologic study and randomized Right Atrial Appendage pacing
  Interventions: Procedure: Pacing RAA study group
- 4. RAA Pacing - control group (Active Comparator): Patients were first submitted to electrophysiological study to assess Delta CTos > or < 50 ms. Then they were randomized to interatrial septum pacing od right atrial appendage. This arm (4) includes patients with Delta CTos <50 ms and randomized Right Atrial Appendage pacing.
  RAA Pacing -Control Group: Patients with Delta CTos <50 ms (control group) at the electrophysiologic study and randomized Right Atrial Appendage pacing
  Interventions: Procedure: Pacing RAA control group

INTERVENTIONS:
Procedure: IAS pacing - study group — site of implant and permanent pacing
  Arms: 1. IAS pacing - study group
Procedure: IAS pacing control group — site of implant and permanent pacing
  Arms: 2. IAS pacing-control group
Procedure: Pacing RAA study group — site of implant and permanent pacing
  Arms: 3. RAA Pacing - study group
Procedure: Pacing RAA control group — site of implant and permanent pacing
  Arms: 4. RAA Pacing - control group

SUMMARY:
This study is a long-term, prospective, and controlled evaluation of the incidence of persistent atrial fibrillation (AF) in patients with severe intra-right atrial conduction delay paced with preventive algorithms at the interatrial septum (IAS) versus right atrial appendage (RAA).

DETAILED DESCRIPTION:
The EPASS is a multicenter, prospective, randomized, and controlled study.

Prior to entering the study, the patient should be informed and provide a written consent. In addition, the patient should meet all selection criteria. The Investigator has to check that all selection criteria are satisfied. Then the patient undergoes pacemaker implantation, receiving a pacemaker model T70 or Selection 9000 (or later version).

Patients eligible for the study are enrolled and submitted to the evaluation of intra-light atrial conduction delay before device implantation. Besides, they are assigned to the group with severe RA conduction delay or with normal conduction delay. The randomization of the pacing site for both groups depends on the value of right atrial conduction delay, together with the associated diseases of the patients, sex and age. After implantation, a stabilization phase of 3-5 weeks is required to stabilize the leads: during this period the physician can optimize the device parameters. Neither the data regarding AF episodes nor cardioversion are collected.

At the end of the stabilization phase the patient undergoes the 1st study follow-up and starts the monitoring period lasting 2 years. Regular follow-ups and data collection are scheduled every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic sinus node dysfunction
* More than 18 years old
* Signed informed consent

Exclusion Criteria:

* Less than 18 years old
* Pregnancy
* Anamnestic transient ischemic attack (TIA) or stroke
* Neoplastic or any other severe disease reducing life expectancy
* Heart surgery in the last 3 months
* Left atrial diameter > 55mm, determined in the parasternal long-axis view (during either sinus rhythm or atrial fibrillation)
* Participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2005-11; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Corbucci, PhD, Study Director — Medtronic; Roberto Verlato, MD, Principal Investigator — Camposampiero Hospital
Locations (8):
- Italy (8):
  - Azienda Ospedaliera di Desenzano del Garda, Desenzano, BS
  - Divisione di Cardiologia, Como, CO
  - Divisione di Cardiologia - CRN, Pisa, PI
  - Divisione di Cardiologia - Ospedale Cisanello, Pisa, PI
  - Divisione di Cardiologia - Ospedale San Pietro Igneo, Fucecchio, Prato
  - Divisione di Cardiologia - Ospedale Molinette, Torino, TO
  - Divisione di Cardiologia - Ospedale Civile ULSS 13, Mirano, VE
  - Divisione di Cardiologia - Presidi Ospedalieri Riuniti, Borgomanero

REFERENCES:
- [Background] Rosenqvist M, Brandt J, Schuller H. Long-term pacing in sinus node disease: effects of stimulation mode on cardiovascular morbidity and mortality. Am Heart J. 1988 Jul;116(1 Pt 1):16-22. doi: 10.1016/0002-8703(88)90244-x. PMID 3394616
- [Background] Stangl K, Seitz K, Wirtzfeld A, Alt E, Blomer H. Differences between atrial single chamber pacing (AAI) and ventricular single chamber pacing (VVI) with respect to prognosis and antiarrhythmic effect in patients with sick sinus syndrome. Pacing Clin Electrophysiol. 1990 Dec;13(12 Pt 2):2080-5. doi: 10.1111/j.1540-8159.1990.tb06946.x. PMID 1704597
- [Background] Santini M, Alexidou G, Ansalone G, Cacciatore G, Cini R, Turitto G. Relation of prognosis in sick sinus syndrome to age, conduction defects and modes of permanent cardiac pacing. Am J Cardiol. 1990 Mar 15;65(11):729-35. doi: 10.1016/0002-9149(90)91379-k. PMID 2316455
- [Background] Sgarbossa EB, Pinski SL, Maloney JD, Simmons TW, Wilkoff BL, Castle LW, Trohman RG. Chronic atrial fibrillation and stroke in paced patients with sick sinus syndrome. Relevance of clinical characteristics and pacing modalities. Circulation. 1993 Sep;88(3):1045-53. doi: 10.1161/01.cir.88.3.1045. PMID 8353866
- [Background] Andersen HR, Nielsen JC, Thomsen PE, Thuesen L, Mortensen PT, Vesterlund T, Pedersen AK. Long-term follow-up of patients from a randomised trial of atrial versus ventricular pacing for sick-sinus syndrome. Lancet. 1997 Oct 25;350(9086):1210-6. doi: 10.1016/S0140-6736(97)03425-9. PMID 9652562
- [Background] Connolly SJ, Kerr CR, Gent M, Roberts RS, Yusuf S, Gillis AM, Sami MH, Talajic M, Tang AS, Klein GJ, Lau C, Newman DM. Effects of physiologic pacing versus ventricular pacing on the risk of stroke and death due to cardiovascular causes. Canadian Trial of Physiologic Pacing Investigators. N Engl J Med. 2000 May 11;342(19):1385-91. doi: 10.1056/NEJM200005113421902. PMID 10805823
- [Background] Attuel P, Pellerin D, Mugica J, Coumel P. DDD pacing: an effective treatment modality for recurrent atrial arrhythmias. Pacing Clin Electrophysiol. 1988 Nov;11(11 Pt 2):1647-54. doi: 10.1111/j.1540-8159.1988.tb06289.x. PMID 2463527
- [Background] 8. Daubert C, Mabo B, Berder V. Arrhythmia prevention by permanent atrial resynchronization in advanced interatrial block. Eur Heart J 1990;11: 237-42.
- [Background] Saksena S, Prakash A, Hill M, Krol RB, Munsif AN, Mathew PP, Mehra R. Prevention of recurrent atrial fibrillation with chronic dual-site right atrial pacing. J Am Coll Cardiol. 1996 Sep;28(3):687-94. doi: 10.1016/0735-1097(96)00232-x. PMID 8772757
- [Background] Delfaut P, Saksena S, Prakash A, Krol RB. Long-term outcome of patients with drug-refractory atrial flutter and fibrillation after single- and dual-site right atrial pacing for arrhythmia prevention. J Am Coll Cardiol. 1998 Dec;32(7):1900-8. doi: 10.1016/s0735-1097(98)00489-6. PMID 9857870
- [Background] 11. Prakash A, Giorgberidze I. Endocardial mapping of sites of conduction delay for atrial premature beats in patients with atrial fibrillation. PACE 1997;20 (part II):1161.
- [Background] Papageorgiou P, Monahan K, Boyle NG, Seifert MJ, Beswick P, Zebede J, Epstein LM, Josephson ME. Site-dependent intra-atrial conduction delay. Relationship to initiation of atrial fibrillation. Circulation. 1996 Aug 1;94(3):384-9. doi: 10.1161/01.cir.94.3.384. PMID 8759080
- [Background] Cosio FG, Palacios J, Vidal JM, Cocina EG, Gomez-Sanchez MA, Tamargo L. Electrophysiologic studies in atrial fibrillation. Slow conduction of premature impulses: a possible manifestation of the background for reentry. Am J Cardiol. 1983 Jan 1;51(1):122-30. doi: 10.1016/s0002-9149(83)80022-8. PMID 6849250
- [Background] Padeletti L, Porciani MC, Michelucci A, Colella A, Ticci P, Vena S, Costoli A, Ciapetti C, Pieragnoli P, Gensini GF. Interatrial septum pacing: a new approach to prevent recurrent atrial fibrillation. J Interv Card Electrophysiol. 1999 Mar;3(1):35-43. doi: 10.1023/a:1009867305678. PMID 10354974
- [Background] Padeletti L, Purerfellner H, Adler SW, Waller TJ, Harvey M, Horvitz L, Holbrook R, Kempen K, Mugglin A, Hettrick DA; Worldwide ASPECT Investigators. Combined efficacy of atrial septal lead placement and atrial pacing algorithms for prevention of paroxysmal atrial tachyarrhythmia. J Cardiovasc Electrophysiol. 2003 Nov;14(11):1189-95. doi: 10.1046/j.1540-8167.2003.03191.x. PMID 14678133
- [Background] Stabile G, Senatore G, De Simone A, Turco P, Coltorti F, Nocerino P, Vitale DF, Chiariello M. Determinants of efficacy of atrial pacing in preventing atrial fibrillation recurrences. J Cardiovasc Electrophysiol. 1999 Jan;10(1):2-9. doi: 10.1111/j.1540-8167.1999.tb00635.x. PMID 9930903
- [Background] De Sisti A, Attuel P, Manot S, Fiorello P, Halimi F, Leclercq JF. Electrophysiological characteristics of the atrium in sinus node dysfunction with and without postpacing atrial fibrillation. Pacing Clin Electrophysiol. 2000 Mar;23(3):303-8. doi: 10.1111/j.1540-8159.2000.tb06753.x. PMID 10750128
- [Background] Leclercq JF, De Sisti A, Fiorello P, Halimi F, Manot S, Attuel P. Is dual site better than single site atrial pacing in the prevention of atrial fibrillation? Pacing Clin Electrophysiol. 2000 Dec;23(12):2101-7. doi: 10.1111/j.1540-8159.2000.tb00783.x. PMID 11202254
- [Background] 19. Attuel P, Pellerin D, Gaston J et al: Latent atrial vulnerability: new means of electrophysiologic investigation in atrial arrhythmias. In Attuel P, Coumel P, Janse M,eds:The Atrium in Health and Disease.Futura Publishing Co.,Inc.,Mt.Kisco,NY,1989,pp159-200.
- [Background] Becker R, Klinkott R, Bauer A, Senges JC, Schreiner KD, Voss F, Kuebler W, Schoels W. Multisite pacing for prevention of atrial tachyarrhythmias: potential mechanisms. J Am Coll Cardiol. 2000 Jun;35(7):1939-46. doi: 10.1016/s0735-1097(00)00631-8. PMID 10841247
- [Background] Duytschaever M, Danse P, Eysbouts S, Allessie M. Is there an optimal pacing site to prevent atrial fibrillation?: an experimental study in the chronically instrumented goat. J Cardiovasc Electrophysiol. 2002 Dec;13(12):1264-71. doi: 10.1046/j.1540-8167.2002.01264.x. PMID 12521344
- [Background] Bailin SJ, Adler S, Giudici M. Prevention of chronic atrial fibrillation by pacing in the region of Bachmann's bundle: results of a multicenter randomized trial. J Cardiovasc Electrophysiol. 2001 Aug;12(8):912-7. doi: 10.1046/j.1540-8167.2001.00912.x. PMID 11513442
- [Background] Hermida JS, Carpentier C, Kubala M, Otmani A, Delonca J, Jarry G, Rey JL. Atrial septal versus atrial appendage pacing: feasibility and effects on atrial conduction, interatrial synchronization, and atrioventricular sequence. Pacing Clin Electrophysiol. 2003 Jan;26(1 Pt 1):26-35. doi: 10.1046/j.1460-9592.2003.00146.x. PMID 12685136
- [Background] Padeletti L, Michelucci A, Pieragnoli P, Colella A, Musilli N. Atrial septal pacing: a new approach to prevent atrial fibrillation. Pacing Clin Electrophysiol. 2004 Jun;27(6 Pt 2):850-4. doi: 10.1111/j.1540-8159.2004.00546.x. PMID 15189515
- [Background] Duytschaever M, Firsovaite V, Colpaert R, Allessie M, Tavernier R. Limited benefit of septal pre-excitation in pace prevention of atrial fibrillation. J Cardiovasc Electrophysiol. 2005 Mar;16(3):269-77. doi: 10.1046/j.1540-8167.2005.40435.x. PMID 15817085
- [Derived] Verlato R, Botto GL, Massa R, Amellone C, Perucca A, Bongiorni MG, Bertaglia E, Ziacchi V, Piacenti M, Del Rosso A, Russo G, Baccillieri MS, Turrini P, Corbucci G. Efficacy of low interatrial septum and right atrial appendage pacing for prevention of permanent atrial fibrillation in patients with sinus node disease: results from the electrophysiology-guided pacing site selection (EPASS) study. Circ Arrhythm Electrophysiol. 2011 Dec;4(6):844-50. doi: 10.1161/CIRCEP.110.957126. Epub 2011 Sep 23. PMID 21946316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment: november 2005 - may 2008 Sites:Ospedale P. Cosma Camposampiero-Ospedale Civile ULSS 13 Mirano-Ospdale Civile,Como-Ospedale Cisanello,Pisa-CRN,Pisa-Ospedale civile, Livorno-Ospedale Molinette, Torino-Presidi Ospedalieri Riuniti,Borgomanero-Ospedale San Pietro Igneo, Fucecchio-Azienda Ospedaliera di Desenzano del Garda Desenzano
Groups:
- IAS Pacing Study Group: Patients with with severe conduction delay (Delta CTos >50 ms, Study Group) randomized to interatrial septum (IAS) pacing.
- IAS Pacing Control Group: Patients without severe conduction delay (Delta CTos <50 ms, Control Group) randomized to interatrial septum (IAS) pacing.
- RAA Pacing Study Group: Patients with severe conduction delay (Delta CTos >50 ms, Study Group) randomized to right atrial appendage (RAA) pacing.
- RAA Pacing Control Group: Patients without severe conduction delay (Delta CTos <50 ms, Control Group) randomized to right atrial appendage (RAA) pacing.
Period: Overall Study
Arm/Group | IAS Pacing Study Group | IAS Pacing Control Group | RAA Pacing Study Group | RAA Pacing Control Group
Started | 30 | 18 | 37 | 17
Completed | 29 | 18 | 36 | 14
Not Completed | 1 | 0 | 1 | 3
Not completed — permAF during stabilization period | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IAS Pacing Study Group | IAS Pacing Control Group | RAA Pacing Study Group | RAA Pacing Control Group | Total
Number analyzed (Participants) | 30 | 18 | 37 | 17 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 8 | 0 | 10
  >=65 years | 28 | 18 | 29 | 17 | 92
Age Continuous [Mean (Standard Deviation); unit: years] | 75 (7) | 79 (6) | 75 (7) | 81 (5) | 77 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 9 | 21 | 10 | 58
  Male | 12 | 9 | 16 | 7 | 44
Region of Enrollment [Number; unit: participants]
  Italy | 30 | 18 | 37 | 17 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Persistent Atrial Fibrillation (AF) After a Mean Follow-up of 15±7 Months: Comparison Between IAS and RAA Pacing in the Study Group
Description: Persistent Atrial Fibrillation (AF) incidence
Time Frame: 1 year
Population: 97 pts completed the study after a mean fu period of 15±7 months.
Measure: Number; unit: Number of patients with persistent AF
Arm/Group | IAS Pacing Study Group | IAS Pacing Control Group | RAA Pacing Study Group | RAA Pacing Control Group
Number analyzed (Participants) | 29 | 18 | 36 | 14
Number of patients with persistent AF | 2 | 2 | 9 | 2
Statistical Analysis 1: Comparison: IAS Pacing Study Group vs RAA Pacing Study Group; Test type: Superiority or Other; p = 0.047, Log Rank; Slope = 3.93

2. Secondary Outcome: Number of Persistent Atrial Fibrillation (AF) Episodes: Comparison Between All Groups
Time Frame: January 2009
Reporting Status: Not Posted

3. Secondary Outcome: Number of Patients With Permanent Atrial Fibrillation (AF)
Time Frame: January 2009
Reporting Status: Not Posted

4. Secondary Outcome: Symptom Scale Questionnaire: Comparison Between All Groups
Time Frame: January 2009
Reporting Status: Not Posted

5. Secondary Outcome: Number of Cardioversion: Comparison Between All Groups
Time Frame: January 2009
Reporting Status: Not Posted

6. Secondary Outcome: Heart Failure: Comparison Between All Groups
Time Frame: January 2009
Reporting Status: Not Posted

7. Secondary Outcome: Time to First Persistent Episode of Atrial Fibrillation (AF)
Time Frame: January 2009
Reporting Status: Not Posted

8. Secondary Outcome: Number of Episodes/Day
Time Frame: January 2009
Reporting Status: Not Posted

9. Secondary Outcome: AF Burden
Time Frame: January 2009
Reporting Status: Not Posted

10. Secondary Outcome: Ventricular Pacing Percentage
Time Frame: January 2009
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | IAS Pacing Study Group | IAS Pacing Control Group | RAA Pacing Study Group | RAA Pacing Control Group
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/18 | 2/36 | 0/14
Other Adverse Events (participants affected / at risk) | 0/29 | 0/18 | 0/36 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IAS Pacing Study Group (N=29) | IAS Pacing Control Group (N=18) | RAA Pacing Study Group (N=36) | RAA Pacing Control Group (N=14)
Hospitalization for HF (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
INVESTIGATOR may publish/present the results of the work. However, INVESTIGATOR shall provide copies of any abstracts, or manuscripts to the sponsor for review at least 30 (thirty) days prior to submittal for publication or presentation. The sponsor shall limit its review to a determination of whether Confidential Information is disclosed and to check for technical correctness. Sponsor shall not attempt to censor or in any way interfere with INVESTIGATOR's presentation or conclusions.